CLINICAL TRIAL: NCT07007806
Title: A Phase 1, Open-Label, Single-Sequence Study to Assess the Effect of Multiple Doses of Omeprazole on the Single-Dose Pharmacokinetics of Bemnifosbuvir/Ruzasvir Fixed-Dose Combination in Healthy Adult Participants
Brief Title: Drug-drug Interaction Study of Omeprazole and Bemnifosbuvir/Ruzasvir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-011
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Omeprazole; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm (n=20) (Experimental)
  Interventions: Drug: Treatment A-Bemnifosbuvir/Ruzasvir FDC administered fasting; Drug: Treatment B-Omeprazole 20 mg dose administered fasting; Drug: Treatment C-Bemnifosbuvir/Ruzasvir FDC administered simultaneously with 20 mg dose of Omeprazole fasting; Drug: Treatment D-Bemnifosbuvir/Ruzasvir FDC administered 0.5 hour prior to 20 mg dose of Omeprazole; Drug: Treatment E-Omeprazole 40 mg administered fasting; Drug: Treatment F-Bemnifosbuvir/Ruzasvir FDC administered 2 hours after 40 mg dose Omeprazole

INTERVENTIONS:
Drug: Treatment A-Bemnifosbuvir/Ruzasvir FDC administered fasting — On day 1 single 550 mg/180 mg dose BEM/RZR FDC (2 × 275 mg/90 mg FDC tablets) will be administered under fasting conditions.
  Other Names: BEM/RZR FDC; BEM (AT-527)/RZR (AT-038)
Drug: Treatment B-Omeprazole 20 mg dose administered fasting — On Day 4 to Day 13, a 20 mg dose omeprazole (1 × 20 mg) will be administered QD under fasting conditions.
  Other Names: Omeprazole; Prilosec®
Drug: Treatment C-Bemnifosbuvir/Ruzasvir FDC administered simultaneously with 20 mg dose of Omeprazole fasting — On Day 8, a single 550 mg/180 mg dose BEM/RZR FDC (2 × 275 mg/90 mg FDC tablets) will be administered under fasting conditions simultaneously with a 20 mg dose omeprazole (1 × 20 mg).
  Other Names: BEM/RZR and Omeprazole; BEM (AT-527)/RZR (AT-038) and Prilosec®
Drug: Treatment D-Bemnifosbuvir/Ruzasvir FDC administered 0.5 hour prior to 20 mg dose of Omeprazole — On Day 13, a single 550 mg/180 mg dose BEM/RZR FDC (2 × 275 mg/90 mg FDC tablets) will be administered 0.5 hour before the administration of a 20 mg dose omeprazole (1 × 20 mg).
  Other Names: BEM/RZR and Omeprazole; BEM (AT-527)/RZR (AT-038) and Prilosec®
Drug: Treatment E-Omeprazole 40 mg administered fasting — On Day 14 to Day 22, a 40 mg dose omeprazole (2 × 20 mg) will be administered QD under fasting conditions.
  Other Names: Omeprazole; Prilosec®
Drug: Treatment F-Bemnifosbuvir/Ruzasvir FDC administered 2 hours after 40 mg dose Omeprazole — On Day 18, a single 550 mg/180 mg dose BEM/RZR FDC (2 × 275 mg/90 mg FDC tablets) will be administered 2 hours after the administration of a 40 mg dose omeprazole (2 × 20 mg).
  Other Names: BEM/RZR and Omeprazole; BEM (AT-527)/RZR (AT-038) and Prilosec®

SUMMARY:
Drug-drug interaction study between Omeprazole and Bemnifosbuvir/Ruzasvir (BEM/RZR)

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use acceptable contraceptive methods through at least 90 days after the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18.5-30 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
PK of BEM/RZR | Day 1, 8, 13, 18
  Cmax
PK of BEM/RZR | Day 1, 7, 8, 13, 18
  AUC
PK of Omeprazole | Day 7, 8
  Cmax
PK of Omeprazole | Day 7, 8
  AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Cypress, California, United States